CLINICAL TRIAL: NCT04909268
Title: PneumoVIH : Prevention of Missed Opportunities for HIV Diagnosis by Promoting HIV Testing of Patients With Pneumococcal Pneumonia at Nice University Hospital
Brief Title: Prevention of Missed Opportunities for HIV Diagnosis by Promoting HIV Testing of Patients With Pneumococcal Pneumonia at Nice University Hospital (PneumoVIH)
Acronym: PneumoVIH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 21Bacterio01
Record Dates: First submitted 2021-05-11; First posted 2021-06-01 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Pneumonia, Pneumococcal; Hiv
MeSH Terms: conditions — Pneumonia, Pneumococcal; Acquired Immunodeficiency Syndrome | interventions — HIV Testing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with positive pneumococcal antigenuria
  Interventions: Diagnostic Test: HIV testing

INTERVENTIONS:
Diagnostic Test: HIV testing — serology for HIV testing

SUMMARY:
According to usual practices, HIV testing should be performed for each patient diagnosed for pneumococcal pneumonia. Unfortunately, in 2018, only 27% of patients were tested for HIV following pneumococcal pneumonia in Nice University Hospital. The aim of PneumoVIH protocol is to promote HIV testing by reminding good practices to physicians. To achieve this, the team of the bacteriology laboratory will contact physicians for each patient positive for pneumococcal antigenuria to suggest HIV testing. This prospective public health action will aim to integrate this HIV test into routine care and to evaluate benefits through the number of HIV positive patients that will be diagnosed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older with validated diagnosis of bacterial pneumococcal pneumonia.

Exclusion Criteria:

* documented history of HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with positive pneumococcal antigenuria
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Testing rate | 1 year
  To evaluate the implementation of the recommendations, HIV testing rate in this population during the study period will be compared with the previous year.

SECONDARY OUTCOMES:
Rate of HIV-positive status discovery | 1 year
  TEvaluating the HIV positivity in patients with bacterial pneumonia or discharged after a visit at the emergency department at the university hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Nice University Hospital, Nice, France

IPD SHARING:
Plan to Share IPD: No
No data sharing is planned